CLINICAL TRIAL: NCT02523885
Title: Descriptive Analysis of Non Steroidal Antiinflammatory Drugs Use in Patients Diagnosed With Community Acquired Pneumonia
Brief Title: Use of Non Steroidal Antiinflammatory Drugs in Patients With Community Acquired Pneumonia
Acronym: ALPAJ
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Professor of Intensive Care Medicine, assistant head of ICU, Hôpital Louis Mourier
Other Study IDs: HLM_JDR3
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Community-acquired Pneumonia
Keywords: Pneumonia, Bacterial [C01.252.620]; Bronchopneumonia [C08.381.677.127]; Pleuropneumonia [C08.730.610.473]; Anti-Inflammatory Agents, Non-Steroidal
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To investigate exposure to nonsteroidal antiinflammatory drugs (NSAIDs) during outpatient management at the early stage of community-acquired pneumonia (CAP) requiring hospital consultation. Non-interventional observational study.

DETAILED DESCRIPTION:
Recent data suggests that such exposure to NSAIDs is associated with delay in CAP diagnosis and antibiotic prescription that influence CAP presention and outcome. The investigators' working hypothesis is that NSAIDs use may mask initial symptoms and delay antimicrobial therapy, thus predisposing to worse outcomes. All patients presenting at one of the three following locations (emergency department, ICU or pneumology ward) with a suspicion of community-acquired pneumonia will be screened for eligibility. Exposure or not to NSAIDs will be investigated. Clinical, biological and radioloigcal features and outcome of CAP will be compared with respect to NSAIDs exposure.

ELIGIBILITY:
Inclusion Criteria: at least two among the following signs

* temperature > 37.8 °C
* respiratory rate > 25/min
* heat rate > 100/min
* cough
* expectoration
* chest pain
* crackles upon lung auscultation

and new infiltrate on the chest x-ray

Exclusion Criteria:

* ongoing pregnancy
* sickle cell disease
* tracheostomy
* long term oxygen therapy
* cystic fibrosis or bronchiectasis
* neutropenia (< 500 cells/mm3)
* ongoing solid or hematologic cancer or anticancerous chemotherapy
* HIV infection
* liver cirrhosis
* long term corticosteroid treatment (20mg per day equivalent prednisone for more than 15 days)
* preexisting treatment with NSAIDs for more than 15 days
* hospital admission for more than 48hours
* aspiration pneumonia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patient presenting either to the emergency department or admitted directly to the ICU or the pneumology ward with a suspicion of CAP will be screened
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
binary composite primary endpoint | 28 days
  presence or absence of one or more of the following : occurrence of at least one pneumonia-related complication; need for ICU admission; prolonged length of hospital stay.
  pneumonia-related complications include: worsening of hypoxemia; need for mechanical ventilation; occurrence or increase of pleural effusion; empyema; occurrence of septic shock;

SECONDARY OUTCOMES:
pneumonia severity index | 2 days
  the pneumonia severity index calculated at inclusion will be compared in exposed and non-exposed to NSAID patients
CURB score at inclusion | 2 days
  the CURB score (confusion, blood urea nitrogen, respiratory rate and systolic blood pressure) at inclusion will be compared in exposed and non-exposed to NSAID patients
duration of antimicrobial therapy | 28 days
occurence of a nosocomial infection | 28 days
  occurrence of nosocomial infections (including nosocomial pneumonia, catheter-related blood stream infection, and urinary tract nosocomial infection) will be compared in exposed and non-exposed to NSAID patients
28-day mortality | 28 days

OTHER OUTCOMES:
chest pain | 2 days
  presence or absence of chest pain at inclusion will compared between exposed and non-exposed to NSAID patients

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien RICARD, MD, PhD, Study Chair — Asssistance Pulique - Hôpitaux de Paris; Muriel FARTOUKH, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Jonathan MESSIKA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Guillaume Voiriot, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; David Hajage, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Louis Mourier Hospital, Colombes
  - Hôpital Max Fourestier, Nanterre
  - Tenon Hospital, Paris

REFERENCES:
- [Background] Voiriot G, Dury S, Parrot A, Mayaud C, Fartoukh M. Nonsteroidal antiinflammatory drugs may affect the presentation and course of community-acquired pneumonia. Chest. 2011 Feb;139(2):387-394. doi: 10.1378/chest.09-3102. Epub 2010 Aug 19. PMID 20724739
- [Background] Messika J, Sztrymf B, Bertrand F, Billard-Pomares T, Barnaud G, Branger C, Dreyfuss D, Ricard JD. Risks of nonsteroidal antiinflammatory drugs in undiagnosed intensive care unit pneumococcal pneumonia: younger and more severely affected patients. J Crit Care. 2014 Oct;29(5):733-8. doi: 10.1016/j.jcrc.2014.05.021. Epub 2014 Jun 4. PMID 24997726